CLINICAL TRIAL: NCT07130669
Title: A Facial Expression-based Personalization Engine (FPE) for Monitoring and Modulating Real-time Effective Engagement in Cognitive Training in Older Adults at Risk for AD/ADRD (CogT FACE Study Phase II)
Brief Title: FACE Phase II (a Stage II Trial)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Feng Lin, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 82182
Record Dates: First submitted 2025-08-05; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: MCI; Subjective Cognitive Decline (SCD); Mild Behavioral Impairment
MeSH Terms: interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- unsupervised cognitive training with personalized engine (Experimental): total 6 week intervention
  Interventions: Behavioral: Cognitive Remediation
- unsupervised cognitive training without personalized engine (Active Comparator)
  Interventions: Behavioral: Cognitive Remediation II

INTERVENTIONS:
Behavioral: Cognitive Remediation — computerized cognitive training with a closed-loop human machine interface that monitor facial expression as engagement status of the person
  Arms: unsupervised cognitive training with personalized engine
Behavioral: Cognitive Remediation II — traditional computerized cognitive training
  Other Names: traditional computerized cognitive training
  Arms: unsupervised cognitive training without personalized engine

SUMMARY:
How to ensure adherence to computerized cognitive training in unsupervised circumstances (e.g., at-home, self-administered) in older adults at risk for Alzheimer's disease (AD) or AD related dementia (AD/ADRD) is understudied. The objective of the R33 study is to test a novel facial expression-based personalization engine (FPE) for monitoring and modulating real-time effective engagement, with an ultimate goal of enhancing long-term adherence in unsupervised cognitive training in older adults at risk for AD/ADRD. Here, Effective engagement is defined as the extent to which someone is actively engaged and performing with significant attention and enjoyment while training, addressing a balance between adherence and cognitive gains/plasticity from the training. Based on previous work, the hypotheses include that (1) mental fatigue revealed in facial expressions will reflect a trainee's degree of effective engagement, which can be modified by modulating task novelty; (2) the proposed FPE will ensure the effective engagement in cognitive training by monitoring trainee facial expressions and modulating training in response, promoting the trainee's long-term adherence to the training and cognitive plasticity. A Stage II intervention efficacy study will be conducted to compare effective engagement and adherence in unsupervised cognitive training between training programs with vs. without FPE in older adults at risk for AD/ADRD. The proposed FPE may assist in monitoring and improving effective engagement and adherence in older adults with unsupervised cognitive training. In the current application, FPE in a cognitive training program called speed of processing training will be tested. However, such FPE may be embedded to any computerized cognitive training in future studies to help address adherence related issues.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking
2. Aged 60-89
3. Living in a home, or independent- or assisted-living facility
4. Adequate visual and hearing acuity
5. Anti-depressants, antipsychotics, and/or anxiolytics have been stable for at least 7 days
6. Memory medications have been stable for at least 3 months
7. Absence of neurological/vascular disorder (For neurological disorders with minor symptoms check with PI on case-by-case basis)

Exclusion Criteria:

1. be enrolled in another intervention study aimed at improving cognition
2. live in nursing home
3. diagnosed with Multiple Sclerosis, TBI, chronic heart failure, Parkinson's disease, dementia

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-31 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
multi-modal effective engagement index (AID) | up to 8 weeks, throughout the intervention sessions
  facial expression+ECG

SECONDARY OUTCOMES:
the time spent on training | up to 8 weeks, throughout the intervention sessions
self-report perceived fatigue | up to 8 weeks, throughout the intervention sessions
  likert scale, 6 items, summarized as 0-10 points
memory | baseline assessment at week 0, post-intervention assessment at week 7, followup assessment at week 13
  BVMT-R delayed recall t score
executive function | baseline assessment at week 0, post-intervention assessment at week 7, followup assessment at week 13
  EXAMINER composite score

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University CogT Lab, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No